CLINICAL TRIAL: NCT05995821
Title: Immunobiology Blood and Tissue Collection of Upper Aerodigestive Malignancies
Status: Recruiting | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Stand Up To Cancer (Other)
Responsible Party: Sponsor
Other Study IDs: J1655; IRB00100653 (Other: Johns Hopkins IRB)
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Cancer; Lung Cancer; Gastrointestinal Cancer
Keywords: Upper Aerodigestive Malignancies; Upper Gastrointestinal (GI) Tract; Thorax; Immunobiology; Immunomodulatory
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Tissue Sample Acquisition:
    * Excess material collected in the course of therapeutic procedures that are clinically indicated; or
    * New biopsies performed for research purposes (e.g., a palpable subcutaneous nodule, or a lymph node that is accessible by ultrasound or computed tomography scan guidance under local anesthesia).
  * Blood Sample Acquisition: A peripheral blood sample will be collected from each participating subject for the isolation and cryopreservation of viable peripheral blood mononuclear cells, serum, and plasma.
  * Leukapheresis: patients may undergo pheresis for the purpose of collecting large numbers of leukocytes for research purposes.
  * Buccal smears
  * Bronchoscopy: Endobronchial brushings +/- biopsies
  * Nasal Epithelium Collection
  * Expectorated Sputum Collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Upper Aerodigestive Malignancies: Patients with cancer of the head and neck, thorax and upper gastrointestinal tract, who are receiving or may receive treatments known or hypothesized to have an immunomodulatory antitumor effect.
  Interventions: Other: Collection of biological specimens

INTERVENTIONS:
Other: Collection of biological specimens — Collection of tumor, blood, lymph nodes, white blood cells, mouth cells (buccal smears) scraped from the inside of your cheek, urine, saliva, or other tissue samples.

SUMMARY:
This research is being done to collect and store biological specimens (biospecimens) from people with cancer, regardless of tumor type, who are receiving treatments known or thought to have an effect on the immune system.

The goal of this discovery and exploratory study is to:

* Understand changes in the immune system associated with various cancer treatments, in order to better design new therapies or tests to predict how these treatments might work.
* Identify risk factors for those who go on to develop side effects from immunotherapy.
* Identify the molecular features associated with response and resistance to cancer therapies and immunotherapy using integrative genomic and immune repertoire characterization.
* Capture and characterize systemic tumor burden by minimally invasive analyses of circulating tumor DNA.

Participants may be asked to:

* Donate samples of tumor, blood, lymph nodes, white blood cells, mouth cells (buccal smears) scraped from the inside of participant's cheek, urine, saliva, or other tissue samples.
* Complete questionnaires about immunotherapy side effects at baseline and with follow-up appointments.
* Undergo knee x-rays.
* Allow the use of demographic and clinical information.

DETAILED DESCRIPTION:
The Immunobiology Blood and Tissue Collection of Upper Aerodigestive Malignancies Protocol is a discovery and exploratory protocol that will enable the investigators to obtain and archive biological specimens from patients with cancer of the head and neck, thorax and upper gastrointestinal tract, who are receiving or may receive treatments known or hypothesized to have an immunomodulatory antitumor effect. The investigators aim to conduct immunologic studies across tumor types and treatment modalities in order to accomplish the following:

1. Gain mechanistic insights into the potential influence of various forms of cancer therapy on antitumor immunity, including but not limited to chemotherapies, kinase inhibitors, angiogenesis inhibitors, immune-modulating monoclonal antibodies, cellular immune therapies and radiation therapy.
2. Define new tumor antigens and the tumor antigens' relevance to disease biology, and correlate antigen expression with immune responses and disease outcomes.
3. Evaluate potential immune-related prognostic or treatment response indicators.
4. Assess the immunologic features of pre-malignant lesions (e.g., atypical or dysplastic nevi, dysplastic bronchial epithelium, colonic adenomas), and compare these features to features of invasive cancers.
5. Investigate the immunobiology of neoadjuvant and adjuvant cancer therapies, including but not limited to cancer vaccines.
6. Develop protein-, RNA-, and DNA-based blood markers to monitor tumor burden and predict and detect tumor relapse.
7. Evaluate the causative mechanisms of immune-related toxicities in patients receiving cancer therapy with immune checkpoint blockade.
8. Characterize factors and molecular pathways in the tumor immune microenvironment that lead to immune suppression, tolerance to tumor antigens, and cancer progression.
9. Understand the epidemiology of and risk factors for particular immune related adverse events (irAEs) including inflammatory arthritis, sicca syndrome and myositis
10. Perform integrative genomic, transcriptomic and immune repertoire characterization of cancers with differential responses to immunotherapy and cancer therapies to determine the molecular features of responding and resistant tumors.
11. Study clonal evolution through genomic, neoantigen, transcriptomic, spatial transcriptomic, and immune repertoire analyses in order to map the evolutionary trajectories of cancer and immune cells under selective pressure of cancer therapies including immune checkpoint blockade.
12. Employ non-invasive molecular assays and analyses of circulating cell-free tumor DNA to capture peripheral tumor and immune compartment dynamics as they relate to response to cancer therapies including immunotherapy.

To support the above research aims, biological specimens obtained and processed in the individual laboratories of the co-investigators will be linked by a centralized demographic database, allowing for the retrieval of information regarding specimen characteristics (e.g., tumor type, treatment exposure, date of specimen retrieval, anatomic site of biopsy, biopsy procedure) and clinical outcomes. Participants starting on immune checkpoint inhibitors will complete a survey when the participants enroll on study to assess for potential risk factors for irAE development. Participants will also undergo knee radiographs to evaluate for osteoarthritis, baseline survey for personal and family historical risk factors, and serial surveys designed to screen for development of irAEs This information will be correlated with the results of exploratory scientific analyses conducted in the laboratories of the co-investigators. Hypotheses generated from this work are expected to support future hypothesis-driven scientific investigations and clinical trial development.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a pathologically confirmed or clinically suspected upper aerodigestive malignancy who may be candidates for known or potentially immunomodulating treatments
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with known significant contraindications for venipuncture (e.g., hemoglobin <8.5 g/dL) will be excluded from the blood collection component of the study
* Patients with known significant contraindications for biopsy (e.g., severe bleeding diathesis) will be excluded from the tissue biopsy component of the study
* Patients with known significant contraindications for bronchoscopy (e.g., airway concerns, significant cardiac disease) will be excluded from the bronchoscopy component of the study
* Unable or unwilling to read English and complete forms/questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both men and women and members of all races and ethnic groups are eligible for participation in this tissue and blood collection protocol. An unlimited number of subjects may be accrued to this study at the Johns Hopkins University.
  Potential research subjects will be identified by their primary physician/clinical team. The research subjects will be patients with cancer of the head and neck, thorax and upper gastrointestinal tract, who are receiving or may receive treatments known or hypothesized to have an immunomodulatory antitumor effect. The immunologic studies will be conducted across tumor types and treatment modalities.
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2016-08-25 (Actual); Primary Completion 2026-08-25 (Estimated); Study Completion 2026-08-25 (Estimated)

PRIMARY OUTCOMES:
Demographic and clinical data obtained via chart review | 10 years
  This is a clinic based registry of cancer therapy data from participants to be collected over time.
Biological specimens obtained from cancer patients | 10 years
  This is a virtual tissue bank containing biological specimens from participants collected over time.

CONTACTS AND LOCATIONS:
Overall Officials: Valsamo Anagnostou, MD, PhD, Principal Investigator — Johns Hopkins University; Joseph Murray, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No